CLINICAL TRIAL: NCT04390841
Title: Clinical Trial for Pre-market Registration of Biotronik Qubic Stim Cardiac Stimulator
Brief Title: Qubic Stim Cardiac Stimulator in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik (Beijing) Medical Device Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EP034
Record Dates: First submitted 2020-02-24; First posted 2020-05-18 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Arrhythmia
Keywords: Paroxysmal supraventricular tachycardia; Ventricular arrhythmia; Atrial fibrillation; Atrial flutter
MeSH Terms: conditions — Arrhythmias, Cardiac; Tachycardia, Ventricular; Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm ( Qubic Stim Cardiac Stimulator ) (Experimental): There is only one Arm in this trial, the subjects who meet the inclusion and exclusion criteria will receive the intracardiac electrophysiological examination, during which the subjects will be subject to diagnostic electrical stimulation by the Qubic Stim Cardiac Stimulator. The subjects will also receive the clinical follow-up visit after cardiac electrical stimulation until they are discharged from the hospital.
  Interventions: Device: Cardiac Stimulator

INTERVENTIONS:
Device: Cardiac Stimulator — The subjects will receive the intracardiac electrophysiological examination, during which the subjects will be subject to diagnostic electrical stimulation by the Qubic Stim Cardiac Stimulator. The subjects will also receive the clinical follow-up visit after cardiac electrical stimulation until they are discharged from the hospital.

SUMMARY:
106 subjects selected from 3 study sites in China are with indications for intracardiac electrophysiological examination. The trial is to prove the clinical effectiveness and safety of Qubic Stim Cardiac Stimulator in Chinese population.

DETAILED DESCRIPTION:
The trial is a multicenter, prospective and single-arm study. 106 appropriate subjects were selected from 3 study sites in China in accordance with the inclusion and exclusion criteria. The subjects consent to participate in the trial and sign the informed consent. The subjects who meet the inclusion and exclusion criteria will receive the intracardiac electrophysiological examination, during which the subjects will be subject to diagnostic electrical stimulation by the Qubic Stim Cardiac Stimulator. The subjects will also receive the clinical follow-up visit after cardiac electrical stimulation until they are discharged from the hospital. The clinical effectiveness and safety of Qubic Stim Cardiac Stimulator in Chinese population were proved by observing the data collected in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Subjects who are willing to participate and sign the informed consent form, and are able to finish the follow-up at the study site.
3. Subjects with an indication of the intracardiac electrophysiological examination(fit one of the following):

   * Paroxysmal supraventricular tachycardia: atrioventricular reentrant tachycardia or atrioventricular node reentrant tachycardia or atrial tachycardia.
   * Ventricular arrhythmia: Premature ventricular contraction or ventricular tachycardia.
   * Atrial fibrillation.
   * Atrial flutter.

Exclusion Criteria:

1. Previous cases of unsuccessful radiofrequency ablation or recurrence
2. Pregnant and/or lactating women
3. Acute or severe systemic infection was present within 7 days prior to the intracardiac electrophysiological examination
4. Liver and kidney functions were obviously abnormal within 7 days prior to the intracardiac electrophysiological examination
5. Obvious bleeding tendency or blood system disease
6. Cancer and terminal disease
7. Combined with severe organic cardiovascular disease
8. Cerebral apoplexy and other cerebrovascular diseases within the past 3 months
9. Thromboembolic disease
10. Subjects who are participating in other interventional clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yifeng Zhou, PHD, Principal Investigator — China-Japan Friendship Hospital
Locations (3):
- China (3):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - TEDA International Cardiovascular Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm ( Qubic Stim Cardiac Stimulator )
Started | 106
Completed | 104
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm ( Qubic Stim Cardiac Stimulator )
Number analyzed (Participants) | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.39 (15.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 60
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: cm] — Population: Height data were not availiable for 34 of the 104 subjects.
  cm
    number analyzed (Participants) | 70
    (all) | 167.61 (9.17)
Weight [Mean (Standard Deviation); unit: kg] — Population: Weight data were not available for 4 of the 104 subjects.
  kg
    number analyzed (Participants) | 100
    (all) | 70.39 (12.87)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: BMI data were not available for 34 of the 104 subjects.
  kg/m^2
    number analyzed (Participants) | 70
    (all) | 25.68 (3.81)

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With Paced Successfully by Programmed Extrastimulation (PES)
Description: The expected clinical effect: the heart is effectively paced by PES at a set rate of stimulation.
  After the release of electrical stimulation, the stimulation signal can produce an effective cardiac pacing wave.
  The asymptotic normal method is an estimator whose limiting distribution is normal when the sample size n increases indefinitely. For example, the sample mean and sample moment are asymptotically normal estimators. Under a wide range of conditions, the maximum likelihood estimators of unknown parameters are asymptotically normal estimators.
  The exact probability method is a statistical test used to determine whether there is a non-random correlation between two variables.
  The asymptotic normal method and the exact probability method were used to estimate the 95% confidence interval of success rate of diagnostic electrical stimulation performed by heart stimulator.
Time Frame: during the procedure
Population: A total of 106 subjects were enrolled in this trial. There were 2 patients excluded from FAS because withdrew informed consent and not complete intracardiac electrophysiological examination with the study device. There remaining 104 patients were included in FAS. In addition, 2 subjects were excluded from PPS because they did not complete all the six required items during the intracardiac electrophysiological examination according to the protocol. Consequently, 102 patients were included in PPS.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Single Arm ( Qubic Stim Cardiac Stimulator )
Number analyzed (Participants) | 104
participants
  Asymptotic normal method on the basis of full analysis set (FAS) | 98 [95 to 100]
  Exact probability method on the basis of full analysis set (FAS) | 98 [93.2 to 99.8]
  Asymptotic normal method on the basis of per protocol set (PPS): number analyzed (Participants) | 102
  Asymptotic normal method on the basis of per protocol set (PPS) | 100 [99.5 to 100]
  Exact probability method on the basis of per protocol set (PPS): number analyzed (Participants) | 102
  Exact probability method on the basis of per protocol set (PPS) | 100 [96.4 to 100]

2. Primary Outcome: High Rate (Burst) Stimulating Successful Rate
Description: Calculate the percentage of subjects who responded successfully to burst stimulation out of the total number of subjects.
Time Frame: during the procedure
Population: A total of 103 subjects were enrolled in this trial and received high-frequency stimulation from the clinical trial device.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm ( Qubic Stim Cardiac Stimulator )
Number analyzed (Participants) | 103
Participants | 103

3. Primary Outcome: Success Rate of Sinus Node Recovery Time (SNRT) Could be Measured.
Description: Calculate the percentage of subjects who had successful sinus node recovery time (SNRT) measurements out of the total number of subjects.
Time Frame: during the procedure
Population: A total of 103 subjects were enrolled in this trial and performed SNRT stimulating by the clinical trial device.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm ( Qubic Stim Cardiac Stimulator )
Number analyzed (Participants) | 103
Participants | 103

4. Secondary Outcome: Serious Device Adverse Events Caused by Cardiac Stimulator
Description: All adverse events shall be recorded throughout the study. However, only the serious adverse events that are definitely, likely or possibly related to Qubic Stim cardiac stimulator will become the basis of SADE event rate. The number of participants with Serious device adverse events caused by cardiac stimulator will be measured and reported.
Time Frame: from the intracardiac electrophysiological examination to discharge, an average of three days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm ( Qubic Stim Cardiac Stimulator )
Number analyzed (Participants) | 104
Participants | 0

ADVERSE EVENTS:
Time Frame: Collect the adverse event data from the time when subjects signed the informed consent form until they were discharged from the hospital, which typically takes an average of 3 days.
Description: Adverse event (AE) refers to any untoward medical occurrence, accident disease or injury, adverse clinical event. All events related to medical device and surgery are included. The symptom occurred due to the existing condition or disease before the enrollment of subjects are not considered to be AE if its frequency of occurrence or severity is not changed.
  The planned examination that doesn't damage the health of subjects, such as regular screening for cancer, is not considered to be AE.
Arm/Group | Single Arm ( Qubic Stim Cardiac Stimulator )
All-Cause Mortality (participants affected / at risk) | 0/104
Serious Adverse Events (participants affected / at risk) | 0/104
Other Adverse Events (participants affected / at risk) | 19/104
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm ( Qubic Stim Cardiac Stimulator ) (N=104)
Intestinal bacteria flora disturbance (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Distention of constipation (General disorders) | 1 (1)
Abnormal liver function (Hepatobiliary disorders) | 2 (2)
Coronary artery atherosclerosis (Cardiac disorders) | 1 (1)
Vomiting and nausea (Gastrointestinal disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Supraventricular premature beats (Cardiac disorders) | 1 (1)
Blood-stained sputum (Blood and lymphatic system disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Dizziness (General disorders) | 3 (3)
Elevated markers of myocardial injury (Cardiac disorders) | 5 (5)
Palpitations (Cardiac disorders) | 1 (1)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Laryngopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Tachycardia sinus (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor has exclusive ownership of the trial data and results. During the clinical trial, the sponsor has the right to access and use all data and results of the trial. Individual clinical trial centers are not allowed to publish and/or report their results until the results of all center are published and/or reported. The sponsor agrees that the leading investigators of the trial will publish the results of the clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT04390841/Prot_SAP_000.pdf